CLINICAL TRIAL: NCT07102251
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HEC-007 Injection After Single-Dose Administration in Healthy Subjects and Multiple-Dose Administration in Overweight or Obese Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, PK/PD of HEC-007 Injection in Healthy and Overweight/Obese Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HEC-007-OB-101
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAD Stage: HEC-007 Injection (Experimental): Administered once
  Interventions: Drug: HEC-007 injection
- SAD Stage: Placebo (Placebo Comparator): Administered once
  Interventions: Drug: Placebo
- MAD Stage: HEC-007 injection (Experimental): Administered for multiple dose
  Interventions: Drug: HEC-007 injection
- MAD Stage: Placebo (Placebo Comparator): Administered for multiple dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HEC-007 injection — Single dose escalation of HEC-007 injection in healthy subjects
  Arms: SAD Stage: HEC-007 Injection
Drug: Placebo — Single dose of placebo in healthy adults
  Arms: SAD Stage: Placebo
Drug: HEC-007 injection — Multiple dose escalation of HEC-007 injection in Overweight or Obese Subjects
  Arms: MAD Stage: HEC-007 injection
Drug: Placebo — Multiple dose of placebo in Overweight or Obese Subjects
  Arms: MAD Stage: Placebo

SUMMARY:
This trial adopts a single-center, randomized, double-blind, placebo-controlled, dose-escalation design to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of HEC-007 Injection after single-dose administration in healthy subjects and multiple-dose administration in overweight or obese subjects.

The trial consists of two parts: Part A is a single ascending dose (SAD) study, planning to enroll 54 Chinese healthy subjects; Part B is a multiple ascending dose (MAD) study, planning to enroll 72 Chinese overweight or obese subjects.

ELIGIBILITY:
Inclusion Criteria:

SAD

1. Subjects understand and comply with the study procedures, voluntarily participate, and sign the informed consent form.
2. Healthy adult subjects (including borderline values) aged 18 to 45 years, regardless of sex.
3. Male subjects weigh no less than 50 kg, and female subjects weigh no less than 45 kg. BMI =Body weight (kg)/height2 (m2), with a body mass index ranging from 19.0 to 35.0 kg/m2 (including boundary values).
4. Normal results or abnormalities deemed clinically insignificant by the investigator in vital signs, physical examination, laboratory tests, electrocardiogram, chest CT, abdominal ultrasound (liver, gallbladder, spleen, pancreas, and both kidneys), and thyroid ultrasound.
5. Female subjects of childbearing potential or male subjects must agree to use effective contraception from signing the informed consent until 6 months after the last administration of the investigational product to avoid pregnancy or impregnating a partner, with no plans for sperm or egg donation or pregnancy.
6. Glycated hemoglobin (HbA1c) <5.7% during the screening period. MAD

1. Subjects understand and comply with the study procedures, voluntarily participate, and sign the informed consent form.

2. Age between 18 to 65 years (inclusive), both male and female. 3. Obesity: BMI ≥28.0 kg/m2; or overweight: 24.0 <BMI <28.0 kg/m2, and with at least one of the following manifestations: prediabetes (as detailed in 14.4), hypertension, dyslipidemia, fatty liver, weight-bearing joint pain, obesity-related dyspnea, or obstructive sleep apnea syndrome.

4. At screening, weight change of < 5% over at least 12 weeks of diet and exercise control alone.

5. Female subjects of childbearing potential or male subjects must agree to use effective contraceptionfrom signing the informed consent until 6 months after the last administration of the investigational product to avoid pregnancy or impregnating a partner, with no plans for sperm or egg donation or pregnancy.

6. Glycated hemoglobin (HbA1c) <6.5% during the screening period.

Exclusion Criteria:

SAD

1. Those diagnosed with type 1, type 2, or other types of diabetes before screening;
2. History or family history of medullary thyroid carcinoma (MTC), thyroid C-cell hyperplasia, or multiple endocrine neoplasia syndrome type 2 (MEN2) during screening, or genetic predisposition to MTC;
3. Acute, chronic, or suspected pancreatitis during screening, or prior pancreatectomy;
4. Those diagnosed with any malignancy within 5 years before screening (except for basal cell carcinoma treated curatively and considered cured);
5. Presence of clinically significant diseases (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immunological, psychiatric, or cardiovascular disorders) during screening;
6. Diseases or conditions affecting gastric emptying or gastrointestinal nutrient absorption during screening;
7. Major surgery within 3 months before screening or planned surgery during the study;
8. History of hypersensitivity to the investigational product or any of its components, or allergic constitution (allergy to two or more drugs or foods).
9. Use of medications (including prescription drugs, over-the-counter drugs, herbal medicines, health supplements, etc.) within 3 months prior to screening that, in the investigator's judgment, significantly affect weight or glucose metabolism;
10. Individuals who have undergone bariatric surgery prior to screening;
11. Those with a history of recurrent skin disorders (e.g., urticaria) or skin lesions at the administration site;
12. Those who received chronic (lasting more than 2 weeks) systemic glucocorticoid therapy (excluding topical, intraocular, intranasal, intra-articular, or inhaled formulations) within 3 months prior to screening, or systemic glucocorticoid therapy within 1 month prior to screening;
13. Female subjects with HbA1c <110 g/L or male subjects with HbA1c <120 g/L at screening, or any other known condition that interferes with HbA1c measurement;
14. Those with suicidal behaviors or ideation within 6 months prior to screening;
15. Use of GLP-1R, GLP-1R/GIPR, GLP-1R/GCGR, or GLP-1R/GIPR/GCGR agonists within 6 months prior to screening;
16. Those with regular alcohol consumption within 3 months prior to screening, defined as more than 14 units of alcohol per week (1 unit = 360 mL beer, 45 mL spirits with 40% alcohol, or 150 mL wine); or those with a positive alcohol breath test during screening; or those unable to comply with the protocol's alcohol restrictions;
17. Those with a history of drug abuse or illicit drug use within 2 years prior to screening, or those with a positive urine drug screen before administration;
18. Smoking more than 5 cigarettes per day within 3 months prior to screening or inability to abstain from smoking during intensive PK blood sampling;
19. Those with a history of needle or blood phobia, intolerance to venipuncture, or difficulty in blood collection;
20. Those with positive results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or Treponema pallidum-specific antibody;
21. Alanine aminotransferase >1.5 × upper limit of normal (ULN), aspartate aminotransferase >1.5 × ULN, alkaline phosphatase >1.5 × ULN, or total bilirubin >1.5 × ULN at screening;
22. Those with blood amylase or lipase > ULN at screening;
23. Those with serum calcitonin ≥20 ng/L at screening;
24. Those with fasting blood glucose ≥6.1 mmol/L or <3.9 mmol/L at screening;
25. Those with glomerular filtration rate (GFR) <90 mL/min/1.73m2 at screening;
26. Fridericia-corrected QT interval (QTcF=QT/RR0.33) >450 ms (for male) or >470 ms (for female) on 12-lead ECG at screening;
27. Use of strong inhibitors or inducers of hepatic metabolic enzymes (CYP1A2, 2A6, 2C8, 2C19, 3A4, and 3A5) within 4 weeks prior to the first dose, including strong inhibitors such as ciprofloxacin, clopidogrel, itraconazole, ketoconazole, ritonavir, troleandomycin, etc., or strong inducers such as rifampin, carbamazepine, phenytoin sodium, St. John's wort, etc.;
28. Use of any prescription drugs, over-the-counter medications, vitamin products, or Chinese herbal medicines within 2 weeks prior to the first dose;
29. Consumption of any foods or beverages affecting CYP3A4, CYP2E1, or CYP2D6 metabolic enzymes, such as grapefruit or grapefruit-containing beverages, within 48 hours prior to the first dose;
30. Ingestion of chocolate, any caffeine-containing or xanthine-rich food or beverage within 48 hours prior to the first dose;
31. Blood donation ≥200 mL, any component blood donation, or total blood loss ≥200 mL due to any reason within 3 months prior to screening, or a history of blood transfusion or blood product use;
32. Participation in other clinical trials within 3 months prior to screening (subjects who withdrew from the study before treatment, i.e., were not randomized or did not receive treatment, may be enrolled in this study);
33. Occurrence of acute illness or concomitant medication use from the signing of the informed consent form until the first dose;
34. Female subjects who are currently breastfeeding or have a positive pregnancy test result at screening;
35. Subjects deemed by the investigator to have other factors unsuitable for participation in this trial.

MAD

1. Those diagnosed with type 1, type 2, or other types of diabetes before screening;
2. Those diagnosed with overweight or obesity caused by other diseases or medications, such as Cushing's syndrome;
3. History or family history of medullary thyroid carcinoma (MTC), thyroid C-cell hyperplasia, or multiple endocrine neoplasia syndrome type 2 (MEN2) during screening, or genetic predisposition to MTC;
4. Acute, chronic, or suspected pancreatitis during screening, or prior pancreatectomy;
5. Those diagnosed with any malignancy within 5 years before screening (except for basal cell carcinoma treated curatively and considered cured);
6. Presence of clinically significant diseases at screening, including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immunological, psychiatric, or cardiovascular disorders (excluding weight-related comorbidities);
7. Any of the following diseases or medical histories within 6 months prior to screening or before randomization: cardiac insufficiency (New York Heart Association [NYHA] Class III or IV), myocardial infarction, unstable angina, uncontrolled arrhythmias requiring treatment (including ventricular tachycardia, ventricular fibrillation, atrial fibrillation, second- to third-degree atrioventricular block, sick sinus syndrome, etc.), coronary artery bypass grafting, percutaneous coronary intervention (diagnostic angiography allowed), cerebrovascular accident (ischemic stroke, hemorrhagic stroke, transient ischemic attack), cirrhosis, etc.;
8. Diseases or conditions affecting gastric emptying or gastrointestinal nutrient absorption during screening;
9. Major surgery within 3 months before screening or planned surgery during the study;
10. History of hypersensitivity to the investigational product or any of its components, or to acetaminophen and its excipients, or allergic constitution (allergy to two or more drugs or foods);
11. Use of medications (including prescription drugs, over-the-counter medications, Chinese herbal medicines, health supplements, etc.) within 3 months prior to screening that, in the investigator's judgment, significantly affect body weight;
12. Subjects taking lipid-lowering or antihypertensive medications with unstable doses within 30 days prior to screening;
13. Individuals who have undergone bariatric surgery prior to screening;
14. Those with a history of recurrent skin disorders (e.g., urticaria) or skin lesions at the administration site;
15. Those who received chronic (lasting more than 2 weeks) systemic glucocorticoid therapy (excluding topical, intraocular, intranasal, intra-articular, or inhaled formulations) within 3 months prior to screening, or systemic glucocorticoid therapy within 1 month prior to screening;
16. Female subjects with HbA1c <110 g/L or male subjects with HbA1c <120 g/L at screening, or any other known condition that interferes with HbA1c measurement;
17. Those with suicidal behaviors or ideation within 6 months prior to screening;
18. History of depression or other psychiatric disorders within 6 months prior to screening;
19. Use of GLP-1R, GLP-1R/GIPR, GLP-1R/GCGR, or GLP-1R/GIPR/GCGR agonists within 6 months prior to screening;
20. Those with regular alcohol consumption within 3 months prior to screening, defined as more than 14 units of alcohol per week (1 unit = 360 mL beer, 45 mL spirits with 40% alcohol, or 150 mL wine); or those with a positive alcohol breath test during screening; or those unable to comply with the protocol's alcohol restrictions;
21. Those with a history of drug abuse or illicit drug use within 2 years prior to screening, or those with a positive urine drug screen before the first dose;
22. Smoking more than 5 cigarettes per day within 3 months prior to screening or inability to abstain from smoking during intensive PK blood sampling;
23. Those with a history of needle or blood phobia, intolerance to venipuncture, or difficulty in blood collection;
24. Resting seated blood pressure at screening: systolic blood pressure >160 mmHg or <90 mmHg, diastolic blood pressure >100 mmHg or <55 mmHg;
25. Heart rate at screening >100 beats per minute or <50 beats per minute;
26. Those with positive results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or Treponema pallidum-specific antibody;
27. Alanine aminotransferase >2 × ULN, aspartate aminotransferase >2 × ULN, alkaline phosphatase >1.5 × ULN, or total bilirubin >1.5 × ULN at screening;
28. Blood amylase or lipase > ULN at screening;
29. Those with serum calcitonin ≥20 ng/L at screening;
30. Fasting triglyceride levels ≥5.6 mmol/L at screening;
31. Fasting blood glucose ≥7.0 mmol/L or <3.9 mmol/L at screening; or OGTT 2-hour ≥11.1 mmol/L;
32. Those with glomerular filtration rate (GFR) <90 mL/min/1.73m2 at screening;
33. Fridericia-corrected QT interval (QTcF=QT/RR0.33) >450 ms (for male) or >470 ms (for female) on 12-lead ECG at screening; or severe arrhythmia (second-degree or higher atrioventricular block, ventricular tachycardia, etc.);
34. Use of strong inhibitors or inducers of hepatic metabolic enzymes (CYP1A2, 2A6, 2C8, 2C19, 3A4, and 3A5) within 4 weeks prior to the first dose, including strong inhibitors such as ciprofloxacin, clopidogrel, itraconazole, ketoconazole, ritonavir, troleandomycin, etc., or strong inducers such as rifampin, carbamazepine, phenytoin sodium, St. John's wort, etc.;
35. Consumption of any foods or beverages affecting CYP3A4, CYP2E1, or CYP2D6 metabolic enzymes, such as grapefruit or grapefruit-containing beverages, within 48 hours prior to the first dose;
36. Ingestion of chocolate, any caffeine-containing or xanthine-rich food or beverage within 48 hours prior to the first dose;
37. Blood donation ≥200 mL, any component blood donation, or total blood loss ≥200 mL due to any reason within 3 months prior to screening, or a history of blood transfusion or blood product use;
38. Participation in other clinical trials within 3 months prior to screening (subjects who withdrew from the study before treatment, i.e., were not randomized or did not receive treatment, may be enrolled in this study);
39. Occurrence of acute illness or concomitant medication use from the signing of the informed consent form until the first dose;
40. Female subjects who are currently breastfeeding or have a positive pregnancy test result at screening;
41. Subjects deemed by the investigator to have other factors unsuitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Screening period up to day 43/day 113
The maximum plasma concentration (Cmax) | Post-dose at day 1 to day 43/day 113
Time to maximum plasma concentration (Tmax) | Post-dose at day 1 to day 43/day 113
Terminal half-life (t1/2) | Post-dose at day 1 to day 43/day 113
Apparent clearance (CL/F) | Post-dose at day 1 to day 43/day 113
Apparent volume of distribution (Vz/F) | Post-dose at day 1 to day 43/day 113
Area Under the PlasmaConcentration-TimeCurve (AUC) of HEC-007 | Post-dose at day 1 to day 43/day 113
Changes from baseline in Body Weight | Baseline period up to day 43/day 113
Changes from baseline in waist circumference | Baseline period up to day 43/day 113
Changes from baseline in Fasting Plasma Glucose | Baseline period up to day 43/day 113
Changes from baseline in Fasting Insulin | Baseline period up to day 43/day 113
Changes from baseline in fasting blood lipids | Baseline period up to day 43/day 113